CLINICAL TRIAL: NCT02682329
Title: Combination of Dental Bleaching Techniques, Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Iberoamericana (Other)
Responsible Party: Principal Investigator, Leandro Feliz, DDS, MEd, Universidad Iberoamericana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dental Bleaching Techniques
Record Dates: First submitted 2016-02-03; First posted 2016-02-15 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Tooth Stain
Keywords: Peroxide
MeSH Terms: conditions — Tooth Discoloration | interventions — Hydrogen Peroxide; Carbamide Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CP 10% + HP 40% (Active Comparator): Carbamide Peroxide 10% + Hydrogen Peroxide 40% were administered to each patient on this group. CP at home and HP at office
  Interventions: Other: Hydrogen Peroxide and Carbamide Peroxide
- CP 15% + HP 40% (Active Comparator): Carbamide Peroxide 15% + Hydrogen Peroxide 40% were administered to each patient on this group.CP at home and HP at office
  Interventions: Other: Hydrogen Peroxide and Carbamide Peroxide
- CP 20% + HP 40% (Active Comparator): Carbamide Peroxide 20% + Hydrogen Peroxide 40% were administered to each patient on this group.CP at home and HP at office
  Interventions: Other: Hydrogen Peroxide and Carbamide Peroxide
- HP 10% + HP 40% (Active Comparator): Hydrogen Peroxide 10% + Hydrogen Peroxide 40% were administered to each patient on this group. HP at Home and HP at office
  Interventions: Other: Hydrogen Peroxide and Hydrogen Peroxide

INTERVENTIONS:
Other: Hydrogen Peroxide and Carbamide Peroxide — Carbamide Peroxide + Hydrogen Peroxide were administered to each patient on this group. HP 10% at home and HP 40% at office
  Arms: CP 10% + HP 40%; CP 15% + HP 40%; CP 20% + HP 40%
Other: Hydrogen Peroxide and Hydrogen Peroxide — Hydrogen Peroxide + Hydrogen Peroxide were administered to each patient on this group. HP at home and HP at office
  Arms: HP 10% + HP 40%

SUMMARY:
To determine the effectiveness of combining different concentrations of hydrogen peroxide and carbamide used during tooth bleaching.

DETAILED DESCRIPTION:
120 patiens over 18 years old.

Design:

Hydrogen peroxide (HP) Carbamide Peroxide (CP)

Group 1: CP 10% + HP 40% Group 2: CP 15% + HP 40% Group 3: CP 20% + HP 40% Group 4: HP 10% + HP 40%

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years old
* Student, teacher or administrative personnel at UNIBE.

Exclusion Criteria:

* Dental Hypersensitivity
* Periodontal disease
* Active caries lesions
* Allergy to latex
* Orthodontic treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in color after the intervention | Two weeks
  The color was taken with conventional hade guide VITA by human observation, with the color range from A to D, each color range with 5 classifications. (Ej. A1, A2, A3, A4, A5)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Feliz-Matos L, Hernandez LM, Abreu N. Dental Bleaching Techniques; Hydrogen-carbamide Peroxides and Light Sources for Activation, an Update. Mini Review Article. Open Dent J. 2015 Jan 6;8:264-8. doi: 10.2174/1874210601408010264. eCollection 2014. PMID 25646134